CLINICAL TRIAL: NCT00006040
Title: Phase I Study of Yttrium-90 Labeled HuM195 Combined With Etoposide as a Conditioning Regimen for Autologous Stem Cell Transplantation in Patients With Advanced Myelodysplastic Syndrome and Refractory Leukemia
Brief Title: Radiolabeled Monoclonal Antibody Therapy and Etoposide Followed by Peripheral Stem Cell Transplantation in Treating Patients With Advanced Myelodysplastic Syndrome or Refractory Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-126; CDR0000068055 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1815
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Filgrastim; Etoposide; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: etoposide
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: yttrium Y 90 monoclonal antibody M195

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate cancer cells and deliver radiation to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of radiation and chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy plus etoposide followed by peripheral stem cell transplantation in treating patients who have advanced myelodysplastic syndrome or refractory leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 humanized monoclonal antibody M195 when combined with etoposide as a preparative regimen for autologous peripheral blood stem cell transplantation in patients with advanced myelodysplastic syndrome or refractory leukemia.
* Determine the qualitative toxicities associated with this regimen in this patient population.
* Assess preliminary information on engraftment following this conditioning regimen in these patients.

OUTLINE: This is a dose escalation study of yttrium Y 90 humanized monoclonal antibody M195 (Y90 MOAB M195).

Patients receive Y90 MOAB M195 IV over 40 minutes once between days -12 to -9 and etoposide IV over several hours on day -3. Peripheral blood stem cells or bone marrow are reinfused on day 0. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 1 until hematopoietic recovery.

Cohorts of 3-6 patients receive escalating doses of Y90 MOAB M195 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose limiting toxicities.

Patients are followed between days 10 and 14 and then monthly for 6 months.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Acute myeloid leukemia
  * Accelerated/blastic phase of a myeloproliferative disorder (i.e., greater than 10% blasts in bone marrow or presence of extramedullary disease)
  * Myelodysplastic syndrome
  * Acute lymphocytic leukemia with expression of CD33

    * Greater than 20% blast population
    * No evidence of CNS disease
* Relapsed after previously achieving complete remission
* Must have previously had peripheral blood stem cells or bone marrow cells harvested and cryopreserved while in remission
* Greater than 25% of bone marrow blasts must be CD33 positive

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* LVEF greater than 50% by ECG or MUGA
* No history of cardiomyopathy or symptomatic congestive heart failure

Pulmonary:

* DLCO at least 50% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* HIV negative
* No other concurrent active malignancy
* No known sensitivity to E. coli derived products

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Maslak, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States